CLINICAL TRIAL: NCT07019376
Title: Investigation of the Effects of Visual Biofeedback-assisted Lumbopelvic Movement Training on Pelvic Proprioception, Pelvic Oscillation, Balance and Core Muscle Endurance in Healthy Sedentary Individuals
Brief Title: Investigation of the Effects of Lumbopelvic Movement Training on Different Parameters in Healthy Sedentary Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Fırat Kara, Principal Investigator, Gazi University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: GAZIU-FTR-FK-001
Record Dates: First submitted 2025-06-01; First posted 2025-06-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Exercise Training
Keywords: proprioception; biofeedback; lumbopelvic; exercise; pelvic sway; balance; endurance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Total of 3 groups including the control group who did not receive any training
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Visual biofeedback supported group (Active Comparator): participants will perform lumbopelvic exercises for 8 weeks, 2 sessions per week for 8 weeks by providing visual biofeedback with a laser.
  Interventions: Other: Visual biofeedback supported lumbopelvic movement training
- Visual biofeedback unsupported group (Active Comparator): Participants will perform lumbopelvic exercises for 8 weeks, 2 sessions per week, without any biofeedback support.
  Interventions: Other: visual biofeedback unsupported lumbopelvic movement training
- Control Group (No Intervention): control group not receiving any exercise

INTERVENTIONS:
Other: Visual biofeedback supported lumbopelvic movement training — 6 exercises that provide movement of the lumbopelvic region will be performed for 8 weeks and 2 times each week. The exercises will be followed visually with the help of a laser.
  Arms: Visual biofeedback supported group
Other: visual biofeedback unsupported lumbopelvic movement training — 6 exercises that provide movement of the lumbopelvic region will be performed for 8 weeks and 2 times each week. The exercises will be the same exercises as the group with laser support, but no visual support will be provided.
  Arms: Visual biofeedback unsupported group

SUMMARY:
The aim of this study was to investigate the effects of visual biofeedback-assisted lumbopelvic movement training on pelvic proprioception, pelvic oscillation, lower extremity static and dynamic balance and core muscle endurance in sedentary healthy individuals.

DETAILED DESCRIPTION:
The lumbopelvic region is an anatomical region where the lumbar spine and pelvis move in harmony in terms of timing and intensity, called the lumbopelvic rhythm, which requires the static, dynamic and neural system to work together, formed by local and global muscles, osteoligamentous structures and neural control. It acts as a force bridge between the lower and upper extremities. Pain, disability, limited activations, atrophy and especially decreases in motor control and proprioception can negatively affect the rhythm and stabilisation in the region. Exercises that contribute to the movement and stabilisation of the lumbopelvic region. There are studies showing that it re-facilitates synaptogenesis, synaptic potentials and reorganisation in areas represented by movement in the motor cortex.

The pelvis makes sinusoidal up-down movements in the frontal and sagittal planes and rotational movements in the transverse plane during walking. These movements are provided by the local and global muscles surrounding the pelvis and hip joint. The reduction of pelvic oscillations in the normal gait pattern may lead to decreased energy expenditure and increased muscle force production.

Lumbopelvic proprioception plays an important role in providing neuromuscular control, creating effective movement, providing coordination, revealing muscle activation at the appropriate timing, preventing spinal and lower extremity injuries and reducing lumbar pain. Decreased proprioceptive sensation leads to impaired movement of the lumbopelvic region and lower and upper extremities, as well as pain and injuries.

In case of weakening of lumbopelvic neuromuscular control and spinal proprioception, significant losses in balance and muscle strength and endurance occur. In order to gain proprioception, balance and strength-endurance parameters should be focused on, and in order to gain balance and strength-endurance parameters, proprioception sense should be developed.

In this direction, the investigators think that lumbopelvic movement training accompanied by visual biofeedback will have a direct effect on pelvic oscillations, lumbar, lumbopelvic, hip and knee proprioception, lower extremity balance and core muscle endurance and these effects will be reflected on the health parameters and daily living activities of individuals. For this purpose, the investigators aim to evaluate the effects of lumbopelvic movement training. At the same time, as a result of the literature review, it is aimed to eliminate the deficiency in this field.

ELIGIBILITY:
Inclusion Criteria:

* sedentary individuals who are not interested in any sport
* individuals without any spine or hip pain problems
* individuals who have not undergone any spine or hip surgery
* individuals who volunteered to participate in the study

Exclusion Criteria:

* athlete individuals who are interested in any sport
* individuals with any spine or hip pain problems
* individuals who have undergone any spine or hip surgery
* individuals who did not volunteered to participate in the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2025-06-04 (Actual); Primary Completion 2025-11-29 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Proprioception | one week
  Proprioception of the lumbopelvic region is evaluated. The movement closest to the target point indicates good proprioception.

SECONDARY OUTCOMES:
Pelvic Sway | one week
  The oscillation of the pelvis will be assessed with an oscillometry device (GYKO) placed at the lumbar 3-5 level. The participant will be asked to walk 10 m and the device will record the oscillation of the pelvis in the anterior-posterior, medial-lateral directions and the total oscillation area during walking.
Balance | one week
  The participant's static and dynamic balance will be measured on the Hurlab Smartbalance device. Functional dynamic balance measurement will be measured with the lower extremity Y balance test.
Core Muscle Endurance | one week
  Evaluation of core muscle endurance will be performed with the Wall Sit Hold, which have proven to be effective in the literature. In the Wall Sit Hold test, individuals will be asked to stand in a squat position with the hip and knee flexed and the back in full contact with the wall and to lift their right or left foot up and wait. The hold time will be recorded in seconds. 3 trials will be made for each foot and the results will be averaged. The higher the data obtained, the higher the core muscle endurance.
Core Muscle Endurance | one week
  In the Trunk Flexion Hold test, the individuals will be asked to sit on their hips and extend their upper body to the feet and knees that are lifted off the floor and wait in this position. The holding time will be recorded in seconds. The hold time will be recorded in seconds. 3 trials will be made for each foot and the results will be averaged. The higher the data obtained, the higher the core muscle endurance.
Core Muscle Endurance | one week
  In the Horizontal Trunk Hold test, individuals will be asked to extend both arms to the side without bending their back and wait in the crawling position. The hold time will be recorded in seconds. 3 trials will be made for each foot and the results will be averaged. The higher the data obtained, the higher the core muscle endurance.

CONTACTS AND LOCATIONS:
Overall Officials: Fırat Kara, Phd Student, Principal Investigator — Nuh Naci Yazgan University
Locations (1):
- Nuh Naci Yazgan University, Kayseri, Kocasinan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No